CLINICAL TRIAL: NCT05120921
Title: OSCAR (Osteopathic Single CAse Research) - Assessing the Effects of Standard and Biopsychosocially-informed Osteopathic Management for Patients With Non-specific Low Back Pain: A Single Case Experimental Design (SCED)
Brief Title: Osteopathic Single CAse Research for Patients With Chronic Low Back Pain
Acronym: OSCAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College of Osteopathy (Other)
Collaborators: Osteopathic Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: OSCAR_LBP
Record Dates: First submitted 2021-10-21; First posted 2021-11-16 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Chronic Low-back Pain
MeSH Terms: interventions — Self-Management; Exercise Therapy

STUDY DESIGN:
Intervention Model Description: The first group of patients will receive standard osteopathic management. The second group will receive biopsychosocially informed osteopathic management.
Who Masked: Outcomes Assessor
Masking Description: The statistician will be blinded to which group patients were allocated to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- standard osteopathic manual treatment (Active Comparator): Pragmatic individualised osteopathic manual treatment which is a system of diagnosis and treatment for a wide range of musculoskeletal conditions. Osteopaths take a detailed case history and perform a thorough clinical examination to help understand the nature of patients' pain and symptoms so that they can arrive at a diagnosis. Practitioners use touch, physical manipulation, stretching and massage to help increase the mobility of joints, to relieve muscle/joint tension and pain. Osteopaths often combine a range of other treatment techniques in their approach, such as rehabilitative exercises, advice about how patients can self-manage their condition and educational approaches to help them understand their pain. Osteopathy is a regulated profession (regulated by the General Osteopathic Council) in the UK
  Interventions: Other: Osteopathic Manual Treatment; Other: Self-management; Other: Reassurance
- biopsychosocially informed osteopathic manual treatment (Active Comparator): As for the active comparator + biopsychosocial management: after having a completed a 8-10 hour e-learning on the biopsychosocial model for the management of low back pain, osteopaths will use the same approaches as in the active comparator group, plus techniques to help patients making sense of their symptoms, to develop patients' self-efficacy, and psychosocial management skills.
  Interventions: Other: Osteopathic Manual Treatment; Other: Self-management; Other: Reassurance; Other: Biopsychosocial management

INTERVENTIONS:
Other: Osteopathic Manual Treatment — includes touch, joint manipulations, stretching and massage
  Other Names: Osteopathic Manipulative Technique
Other: Self-management — Providing rehabilitative exercises to patients to do at home
  Other Names: Therapeutic exercises
Other: Reassurance — Reassuring patients on their symptoms, diagnosis and prognosis.
  Other Names: cognitive reassurance; affective reassurance
Other: Biopsychosocial management — Giving a central place to the patient in the decision-making to help them to get back to valued activities.
  Other Names: Enactive approach
  Arms: biopsychosocially informed osteopathic manual treatment

SUMMARY:
This study aims to collect primary data from patients with low back pain to assess the effect of standard osteopathic management and biopsychosocially-informed osteopathic care using a Single-Case Experimental Design.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all osteopaths and patient participants giving written consent will be screened for eligibility. When entering the trial, patients will be randomised to early, intermediate or late intervention with either standard osteopathic management or biopsychosocially-informed osteopathic management.

ELIGIBILITY:
Inclusion Criteria:

* 18 or more years old
* agree to take part in the study and provide formal online consent after having been assessed as capable of providing informed consent by the osteopath
* Being fluent enough in English to be able to understand content of consent forms (and participate in osteopathic treatment without an interpreter)
* Presenting with non-specific low back pain of a duration of a minimum of 12 weeks)
* NRS score between 5 and 9 on a 11-point scale
* PSFS score between 2 and 7 at baseline
* Who can be contacted by email
* Available for an appointment within two days around the randomisation date

Exclusion Criteria:

* Under 18
* Lacking capacity to give consent
* Presenting with low back pain with a known or suspected pathological cause (e.g. infection, cancer or fracture)
* People for whom osteopathic treatment may be contra-indicated (as assessed by the osteopath in the initial consultation) or who disclose information during their course of treatment which requires referral for other medical investigations or care
* LBP of less than 12 weeks
* NRS score below 5 or above 9
* PSFS score above below 2 or above 7
* Patients providing less than 3 data points during baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale changes during the treatment phase (max 6 weeks) and follow-up period (12 weeks) | Up to 18 weeks
  11-item unidimensional measure of pain intensity. The Initiative on Methods, Measurement, and Pain Assessment in Clinical Trials recommendations will be used, i.e. patients will be presented with the numbers from 0 to 10, with 0 meaning 'No pain' and '10' meaning 'Pain as bad as you can imagine,' accompanied by the instructions "Please rate your pain by indicating the number that best describes your pain on average in the last 24h". NPRS is an acceptable measure but should not be used on its own as patients with chronic pain find it does not capture the complexity of their pain experience. It has a high test-retest reliability and a good validity. Patients will be asked to complete the NPRS every day, taking approx. 1 min.
The Patient Specific Functional Scale changes during the treatment phase (max 6 weeks) and follow-up period (12 weeks) | Up to 18 weeks
  PSFS measures functional change in patients with musculoskeletal disorders. Patients choose to list up to 5 activities that they have difficulty with or are unable to perform. They will be asked to continue recording data for the originally chosen activities but can add extra activities if goals change (e.g. due to improving or worsening symptoms). Patients will rate current level of difficulty for each activity on an 11-point scale, where 0 = unable to perform and 10 = able to perform at previous level. Mean averages are calculated by summing the difficulty ratings and dividing by the number of activities. The PSFS is reliable and responsive for patients with chronic low back pain and a Minimum Detectable Change (MDC) is considered to be 3 points for 1 activity or 2 points for the average of 2 or more activities.

SECONDARY OUTCOMES:
Measure Your Medical Outcome Profile 2 | Up to 18 weeks
  MYMOP2 is a self-report questionnaire that lists one or two symptoms and one activity affected by the patient's condition. The first activity the patient participant created in PSFS will automatically be entered into the text of MYMOP2. The follow-up questionnaire is shorter but allows addition of a third symptom. MYMOP2 is a validated, sensitive and responsive outcome measure. A minimum clinically important change (MCIC) in score should be between 0.5-1.0, and any change greater than 1.0 is considered clinically significant. Patients will be asked to complete MYMOP2 once a week, taking approx. 5 min.
The Arthritis Research UK Musculoskeletal Health Questionnaire | Up to 18 weeks
  MSK-HQ captures generalised health outcomes that are relevant to patients with a range of musculoskeletal conditions. It achieves high completion rates, excellent test-retest reliability, and has strong convergent validity with reference standards. It includes 14 questions scored on a 0-4 scale (range 0-56, where a higher total score represents better health). A licence has been requested to use the questionnaire online from Oxford University Innovation centre for free. Patients will be asked to complete the MSK-HQ three times, taking approx. 2 minutes.
The Depression, Anxiety, and Positive Outlook Scale | Up to 18 weeks
  DAPOS is a self-administered questionnaire that measures distress and positive affect in chronic musculoskeletal pain populations. It has 11 items: 5 on depression, 3 on positive affect and 3 on anxiety; all answered with a 5-point Likert scale response (ranging from 'almost never' to 'almost all the time'). It has an excellent internal consistency and construct validity in comparison with a variety of measures (SF-36; Pain Catastrophizing Scale; Zung Depression) and an acceptable responsiveness.
The Pain Attitudes and Beliefs Scale (for the osteopaths) | 6 months
  PABS is a 19-item questionnaire with six-point response scales. The questionnaire aims to assess two treatment orientations towards LBP: 'biomedical', where disability and pain are consequences of speciﬁc tissue pathology and treatment aims to treat pathology; and 'behavioural', where practitioners believe in a BPS model of disease, in which pain does not have to be a sign of tissue damage and can be inﬂuenced by social and psychological factors. There is evidence for content and construct validity, internal consistency, reliability and responsiveness. The modified version of the PABS will be used in this project (Cronbach's α Biomedical domain 0.84; Cronbach's α behavioural domain is 0.68).

OTHER OUTCOMES:
Survey about experience of osteopathic treatment and of participating in the SCED study (for patients) | 6 weeks
  At the end of their course of treatment, patients will be asked to complete a final. This questionnaire has been adapted from the Patient Enablement Index for Back Pain and contains 12 questions to assess patients' perceptions of shared decisions making, treatment outcomes, relevance of the measures and acceptability of the data collection processes.
Prognostic surveys (for the osteopaths) | 6 weeks
  Osteopaths will fill in two surveys, one after the initial visit of a patient and one 6 weeks later. It was previously used to assess physical therapists' ability to accurately prognose their patients.
Survey of SCED feasibility and acceptability and impact of the e-learning course on patient care (for the osteopaths) | 9 months
  It was adapted from the Patient Enablement Index. It consists of 12 questions with 11-point Likert scale response options for agreement and satisfaction and 2 open text questions about osteopaths' experiences of SCED processes and outcomes to guide future training and research, taking approx. 5 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Jerry RF Draper-Rodi, D.Prof.(Ost), Principal Investigator — University College of Osteopathy
Locations (1):
- University College of Osteopathy, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Dataset will be made available with the publication or by email request to the PI
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From publication of the results and up to 6 years after trial completion.
Access Criteria: Researchers who provide a methodologically sound proposal. Proposals should be directed to jerry.draper-rodi@uco.ac.uk To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Draper-Rodi J, Vogel S, Bishop A. Effects of an e-learning programme on osteopaths' back pain attitudes: a mixed methods feasibility study. Pilot Feasibility Stud. 2021 Sep 13;7(1):174. doi: 10.1186/s40814-021-00901-4. PMID 34517916
- [Background] Draper-Rodi, J., Vogel, S. and Bishop, A., 2018. Design and development of an e-learning programme: An illustrative commentary. International Journal of Osteopathic Medicine, 29, pp.36-40.